CLINICAL TRIAL: NCT06622954
Title: Protein and Calorie Restriction as Treatment for Prevention of Cardiotoxicity in Women Receiving Chemotherapy.
Brief Title: Dietary Restriction to Prevent Cardiotoxicity in Breast Cancer Patients
Acronym: PROTECT-COR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Franny Jongbloed, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEC-2022-0823
Record Dates: First submitted 2023-09-06; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Cardiotoxicity; Breast Cancer
Keywords: Dietary restriction; Diet; Anthracyclines; High sensitivity troponin T; HsTnT; Oxidative stress; Breast cancer; Cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms | interventions — Proteins

STUDY DESIGN:
Intervention Model Description: Two groups, 1 control group and 1 intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein- and Calorie restriction group (Other): This group will receive the dietary intervention.
  Interventions: Other: Protein- and Calorie restriction
- Control Group (No Intervention): This group will not receive any intervention.

INTERVENTIONS:
Other: Protein- and Calorie restriction — The intervention consists of 30% calorie and 70% protein restriction, based on their daily nutritional intake. The protein and calorie restriction will be given in the form of Scandishake from Nutricia. These are ready available and easy to tailor to the caloric and protein need of each individual study subject.
  Arms: Protein- and Calorie restriction group

SUMMARY:
The goal of this clinical trial is to compare a dietary intervention with a regular diet in patients with early breast cancer undergoing anthracycline based chemotherapy. The main question it aims to answer is:

What are the effects of a short-term diet with 30% caloric and 70% protein restriction (PCR) on cardiotoxicity induced by anthracycline treatment in women with newly diagnosed invasive breast cancer.

Researchers will compare the control group with dietary intervention group to see if cardiotoxicity -measured by concentrations of high-sensitivity troponin T (hsTnT) levels- will be different between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* women with newly diagnosed triple negative breast cancer with an indication for (neo-)adjuvant ATC-based chemotherapy and of intent to start anticancer treatment;
* age between 18 and 75 years;
* written informed consent;
* body mass index ≥ 19.

Exclusion Criteria:

* Allergic to any of the ingredients of the diet;
* Known history of cardiac dysfunction;
* Severe morbidity with the inability to receive anticancer treatment.
* Participation in another clinical trial with an intervention arm (database and/or biobank studies excluded);
* Pregnant women
* Previous treatment with anthracycline
* Estrogen receptor positive status

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
High-sensitivity troponin T (hsTnT) | Bloodsamples will be taken before and 1 hour after each anthracycline based chemotherapy cycle. The cycles are given once every 2 weeks, for 4 cycles in total.
  Cardiotoxicity as determined by the difference in concentrations of high-sensitivity troponin T (hsTnT) levels after protein and calorie restriction and anthracycline treatment in one cycle, delta HsTnT (Δ HsTnT).

SECONDARY OUTCOMES:
Left ventricular ejection fraction and global longitudinal (LVEF and GLS) | 6 months and 12 months after start of anthracycline therapy
  Echocardiography assessment of LVEF and GLS, to evaluate the overall effect on markers of cardiotoxicity and cardiac function.
Creatine kinase | Bloodsamples will be taken before and 1 hour after each anthracycline cycle. The cycles are given once every 2 weeks, for 4 cycles in total.
  Increase in creatine kinase after each cycle
Effect of dietary intervention on tumor volume/response | After chemotherapy cycle 3 or cycle 4 (chemotherapy is given every 2 weeks)
  Radiographic response rate (measured as Complete Response / Partial Response / Stable Disease / Progression of disease, via RECIST method.
Metabolic parameters | Bloodsamples will be taken before and 1 hour after each anthracycline based chemotherapy cycle. The cycles are given once every 2 weeks, for 4 cycles in total.
  Retinol binding protein, albumin and lipid profile.
Other anthracycline-related toxicities | After each anthracycline based chemotherapy cycle, which is given every 2 weeks. There will be 4 cycles in total.
  Measured with CTCAE grading, part of standard of care.
Effect of dietary intervention on pharmacokinetics of anthracycline | Bloodsamples will be taken before and 1 hours after each anthracycline based chemotherapy cycle. The cycles are given once every 2 weeks, for 4 cycles in total.
  Effect of dietary intervention on pharmacokinetics of the anthracycline, as measured by concentrations of anthracycline after each chemotherapy cycle.
Troponin levels | Bloodsamples will be taken before and 1 hour after each anthracycline based chemotherapy cycle. The cycles are given once every 2 weeks, for 4 cycles.
  Difference in troponin levels, before and after each of the other chemotherapy cycles (that are not taken for primary outcome measure), Δ HsTnT.
Brain natriuretic peptide (NT-proBNP) | Bloodsamples will be taken before and 1 hour after each anthracycline based chemotherapy cycle. The cycles are given once every 2 weeks, for 4 cycles in total.
  Increase in brain natriuretic peptide after each cycle
Subjective wellbeing | During each anthracycline chemotherapy cycle. The chemotherapy is given every 2 weeks, in total 4 cycles. Then 6 months and 12 months after start of anthracycline therapy questionnaires will be taken again.
  Subjective wellbeing will be measured using the following questionnaires: EuroQol, VAS-scores, multidimensional fatigue index.

CONTACTS AND LOCATIONS:
Overall Officials: Franny Jongbloed, MD/PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands